CLINICAL TRIAL: NCT04927091
Title: Integrating Addiction Treatment and HIV Services Into Primary Care Clinics in Ukraine
Acronym: IMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Ukrainian Institute on Public Health Policy (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2000020067; 1R01DA043125-01 (NIH)
Record Dates: First submitted 2021-06-10; First posted 2021-06-15 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Hiv; Opioid-use Disorder
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Opioid-Related Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Specialty Addiction Clinic (No Intervention)
- ECHO-IC/QI-enhanced primary care clinic (Experimental)
  Interventions: Other: Integration of HIV and PWID services
- ECHO-IC/QI-enhanced primary care clinic with Pay for Performance (Active Comparator)
  Interventions: Other: Integration of HIV and PWID services

INTERVENTIONS:
Other: Integration of HIV and PWID services — Co-location of clinical services for HIV and PWID patients
  Arms: ECHO-IC/QI-enhanced primary care clinic; ECHO-IC/QI-enhanced primary care clinic with Pay for Performance

SUMMARY:
A randomized controlled trial to:

1. To compare both primary (composite quality health indicator (QHI) scores) and secondary (individual HIV/methadone maintenance treatment (MMT)/TB/primary care QHI scores, quality of life, and stigma) outcomes in an anticipated 1,350 people who inject drugs (PWID) receiving MMT from 13 regions (clusters) and 39 clinical settings using a stratified, phase-in, controlled design over 24 months. After stratifying PWIDs based on their current receipt of MMT, they will be randomized to receive MMT in specialty addiction clinics (N=450) or in an ECHO-IC/QI-enhanced primary care clinic with (N=450) or without (N=450) pay for performance (P4P) incentives.
2. Using a multi-level implementation science framework, to examine the contribution of client, clinician and organizational factors that contribute to the comprehensive composite (primary outcome) and individual (secondary) QHI scores.

DETAILED DESCRIPTION:
Original outcomes were edited and Implementation outcomes were added November 2023.

ELIGIBILITY:
Inclusion Criteria:

* PWID
* Interested in MMT
* Meets DSM-V criteria for Opioid Dependence

Exclusion Criteria:

* Not willing to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1458 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Average percentage of recommended Quality Health Indicator services accessed by participants to assess efficacy | every 6 months up to 24 months
  The total average percentage of the 17 recommended Quality Health Indicator screenings and services that were accessed by participants to assess efficacy. Recommended QHI screenings are as follows: General medical examination; blood analysis; urine analysis; cardiogram; mammogram; cervical cancer screening; prostate cancer screening; hepatitis B screening; hepatitis C screening; HIV screening; CD4 or viral load; ART treatment; TB screening; TB treatment; received take-home MMT; adequate MMT dose; on MMT for 12 months.

SECONDARY OUTCOMES:
Average percentage of recommended HIV Quality Health Indicator services accessed to assess efficacy | every 6 months up to 24 months
  The total average percentage of the 3 HIV Quality Health Indicator screenings and services that were accessed by participants to assess efficacy. Recommended QHI screenings are as follows: HIV screening; CD4 or viral load; ART treatment.
Average percentage of recommended MMT Quality Health Indicator services accessed to assess efficacy | every 6 months up to 24 months
  The total average percentage of the 3 HIV Quality Health Indicator screenings and services that were accessed by participants to assess efficacy. Recommended QHI screenings are as follows: received take-home MMT; adequate MMT dose; on MMT for 12 months.
Average percentage of recommended TB Quality Health Indicator services accessed to assess efficacy | every 6 months up to 24 months
  The total average percentage of the 2 HIV Quality Health Indicator screenings and services that were accessed by participants to assess efficacy. Recommended QHI screenings are as follows: TB screening; TB treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Altice, MD, Principal Investigator — Yale University
Locations (1):
- European Institute for Public Health Policy, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Machavariani E, Esserman D, Dumchev K, Filippovych M, Pykalo I, Ivasiy R, Madden LM, Bromberg DJ, Haddad M, Morozova O, Oliveros D, Ahmad B, Dvoriak S, Altice FL. Integrating Methadone Services Into Primary Care in Ukraine: Two-Year Outcomes From a Randomized Trial. Ann Intern Med. 2025 Dec 9. doi: 10.7326/ANNALS-25-01764. Online ahead of print. PMID 41359964
- [Derived] Pashchenko O, Bromberg DJ, Dumchev K, LaMonaca K, Pykalo I, Filippovych M, Esserman D, Polonsky M, Galvez de Leon SJ, Morozova O, Dvoriak S, Altice FL. Preliminary analysis of self-reported quality health indicators of patients on opioid agonist therapy at specialty and primary care clinics in Ukraine: A randomized control trial. PLOS Glob Public Health. 2022 Nov 2;2(11):e0000344. doi: 10.1371/journal.pgph.0000344. eCollection 2022. PMID 36962514